CLINICAL TRIAL: NCT06023004
Title: Circulating Tumor DNA Guided vs Opportunistic Colonoscopy Screening for CRC Detection After Acute Colonic Diverticulitis - the Diverticulitis Study
Brief Title: The Diverticulitis Study
Status: Active, not recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Odense University Hospital (Other); Regionshospitalet Horsens (Other); University of Southern Denmark (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: The Diverticulitis study
Record Dates: First submitted 2023-08-28; First posted 2023-09-05 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Colonic Diverticulitis; Colorectal Cancer; Acute Diverticulitis
MeSH Terms: conditions — Diverticulitis, Colonic; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — From each patient, blood will be collected between 2 and 6 weeks after the diagnosis of diverticulitis. The blood will be collected before initiation of the bowel cleansing associated with the CRC screening colonoscopy.
  Blood draw: 80 mL - 7 x EDTA tubes, 1 x serum tube
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Controls: Patients diagnosed with diverticulitis through CT scan and scheduled for a colonoscopy. The colonoscopy must result in no detection of colorectal cancer.
- Cases: Patients diagnosed with CRC immediately after an episode of diverticulitis.

SUMMARY:
Acute colonic diverticulitis is when a part of the colon gets swollen and inflamed. The diagnosis is based on a CT scan, which can show thickening of the colonic walls and infiltration of the diverticula. These changes and the concomitant symptoms can overlap with colorectal cancer (CRC). Therefore, the guidelines suggest that people with diverticulitis should be offered a colonoscopy to ensure, that CRC is not the underlying cause of the changes and symptoms.

In Denmark, a lot of people get hospitalized each year due to diverticulitis, and many of them end up having colonoscopies with the purpose of excluding CRC. Currently, there are no methods for guiding colonoscopies following a diverticulitis episode, resulting in numerous unnecessary colonoscopies each year.

In the Diverticulitis study, we want to investigate if a simple blood test analyzed for the presence of circulating tumor DNA (ctDNA), can help us decide who needs a colonoscopy. We will collect blood samples from 220 people with diverticulitis and categorize them into ctDNA positive and negative groups. The ctDNA category will be compared to the colonoscopy results to see if there is a correlation between being ctDNA positive and having a CRC diagnosed at the colonoscopy.

This study could change clinical practice since we anticipate that ctDNA-guided triaging of diverticulitis patients is a cost-effective strategy for selecting diverticulitis patients needing colonoscopy, ensuring detection of the underlying CRC, and significantly reducing the number of patients undergoing unnecessary colonoscopy.

DETAILED DESCRIPTION:
KEY POINTS

* Colonoscopy is recommended after acute diverticulitis to rule out CRC, and yearly more than 2000 colonoscopies are performed.
* CRC incidence is low in the diverticulitis population and most colonoscopies are unnecessary. It takes approximately 100-200 colonoscopies to diagnose just 1 CRC.
* ctDNA is a minimally invasive and extraordinarily powerful biomarker of cancer.

GOALS

● To use ctDNA analysis to triage diverticulitis patients for colonoscopy. Diagnosing the same CRCs, but minimizing the number of patients needing colonoscopy

PERSPECTIVES

* Practice-changing evidence for ctDNA-guided triaging of diverticulitis patients for colonoscopy, an important and well-recognized clinical dilemma in the management of CRC.
* Evaluation of the cost-effectiveness of ctDNA-guided triaging versus standard-of-care.

PROJECT DESCRIPTION For patients who have experienced an episode of acute colonic diverticulitis, Danish and international guidelines recommend opportunistic screening with colonoscopy to rule out CRC as the underlying reason for the diverticulitis symptoms. In Denmark, there are more than 4000 hospitalizations per year due to diverticulitis. Accordingly, a substantial number of post-diverticulitis colonoscopies are performed each year to rule out underlying CRC. Colonoscopy is an invasive procedure associated with discomfort and pain in more than 50% of patients. The procedure also carries the risk of complications such as perforation and hemorrhage, particularly for patients with diseased intestines such as diverticulitis patients. CRC prevalence in suspected diverticulitis patients is low, <2% overall, and as low as 0.5% for uncomplicated diverticulitis. Thus, an unreasonably high number of colonoscopies, ranging from 50 and up to more than 200, are needed to diagnose 1 CRC. In comparison, a >4% CRC prevalence is considered the minimal acceptable among patients selected for follow-up colonoscopy in the Danish nationwide CRC screening program, corresponding to less than 25 colonoscopies per CRC. Hence, it may be questioned whether the current guidelines on follow-up colonoscopy after diverticulitis are at all acceptable, both from a patient perspective and from a health-economy perspective. However, it has been very difficult to change. Consequently, there is an urgent need for a highly sensitive, low-risk, minimally invasive cancer detection test that can be used to triage newly diagnosed diverticulitis patients and ensure that underlying CRC is still diagnosed while minimizing the number of patients needing colonoscopy. Here, we propose to conduct a case/control study to explore the feasibility of using our recently developed TriMeth ctDNA analysis test for this purpose.

We hypothesize that ctDNA analysis can triage diverticulitis patients for colonoscopy and achieve a diagnosis of prevalent CRC but at a substantially lower colonoscopy/CRC ratio. For this purpose, we will use our tumor-agnostic ctDNA analysis "TriMeth". TriMeth was originally developed as a CRC screening tool for selecting individuals from the average-risk population for colonoscopy. Accordingly, the threshold for calling the test positive was set with the objective of high specificity. At 99% specificity, it has a sensitivity of 85%. Based on data from the original development and validation cohorts (400 CRC and 800 controls), we will tailor TriMeth for this specific purpose, i.e., setting the threshold for test positivity to achieve near 100% sensitivity by accepting a lower specificity. Second, we will conduct a case-control study to validate this new TriMeth-diverticulitis threshold in the target population. We expect a minimum of 20 cases with CRC diagnosed at colonoscopy after suspected diverticulitis to be identified through the IMPROVE study (NCT03637686). For each case, 10 controls will be randomly selected (to a minimum of 200 total) from patients with CT-verified diverticulitis and a follow-up colonoscopy without CRC. Diverticulitis patients may at the time of colonoscopy exhibit symptoms, that would in any case serve as an absolute indication for colonoscopy (patients age >40 with changes in bowel habits >1 month, rectal bleeding, iron-deficiency anemia, or excessive weight-loss). Therefore, in addition to blood sampling, we will at the time of CRC diagnosis or negative colonoscopy collect information on other established indicators for colonoscopy. As part of the study, we will conduct a health-economy assessment comparing the TriMeth-guided approach to the current practice of "colonoscopy for all". The primary outcome is the sensitivity and specificity of TriMeth for CRC detection in this population. The secondary outcome is health economy, considering the other indicators for colonoscopy. If high sensitivity and clinically and economically relevant colonoscopy-sparing potential is demonstrated, the data will be presented to the Danish Colorectal Cancer Group and the Danish Health Technology Council with the aim of obtaining approval to change the national guideline and implement the approach.

ELIGIBILITY:
Inclusion Criteria:

* CT-verified diverticulitis eligible for a follow-up colonoscopy

Exclusion Criteria:

* Unable to provide oral and written informed consent
* Recent colonic imaging and no need for renewed visualization of the colonic mucosa deemed by the attending doctor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly CT-verified diverticulitis will be identified by the attending physician at the recruiting surgical departments. Patients fulfilling the inclusion criteria are approached and invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
ctDNA analysis | After recruitment of the last patient, we expect that ctDNA analyses can be performed within 6 months
  Blood samples will be categorized as either ctDNA positive or negative

SECONDARY OUTCOMES:
Cost-effectiveness of treatment | After recruitment of the last patient, we expect that cost-effectiveness analyses can be performed within 12 months
  Assessment of the cost-effectiveness of "ctDNA guided" versus "opportunistic" colonoscopy screening of the diverticulitis patients

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bjørsum-Meyer, MD, PhD, Principal Investigator — Odense University Hospital; Per V Andersen, MD, PhD, Principal Investigator — Odense University Hospital; Kåre A Gotschalck, MD, PhD, Principal Investigator — Regionshospitalet Horsens; Liza Sopina, PhD, Principal Investigator — University of Southern Denmark
Locations (5):
- Denmark (5):
  - Herlev Hospital, Herlev, Capital Region of Denmark
  - Regional Hospital Horsens, Horsens, Central Jutland
  - Regional Hospital Randers, Randers, Central Jutland
  - Regional Hospital Viborg, Viborg, Central Jutland
  - Odense University Hospital, Odense, The Region of Southern Denmark

REFERENCES:
- [Background] Andersen JC, Bundgaard L, Elbrond H, Laurberg S, Walker LR, Stovring J; Danish Surgical Society. Danish national guidelines for treatment of diverticular disease. Dan Med J. 2012 May;59(5):C4453. PMID 22549495
- [Background] Meyer J, Orci LA, Combescure C, Balaphas A, Morel P, Buchs NC, Ris F. Risk of Colorectal Cancer in Patients With Acute Diverticulitis: A Systematic Review and Meta-analysis of Observational Studies. Clin Gastroenterol Hepatol. 2019 Jul;17(8):1448-1456.e17. doi: 10.1016/j.cgh.2018.07.031. Epub 2018 Jul 26. PMID 30056181
- [Background] Jensen SO, Ogaard N, Orntoft MW, Rasmussen MH, Bramsen JB, Kristensen H, Mouritzen P, Madsen MR, Madsen AH, Sunesen KG, Iversen LH, Laurberg S, Christensen IJ, Nielsen HJ, Andersen CL. Novel DNA methylation biomarkers show high sensitivity and specificity for blood-based detection of colorectal cancer-a clinical biomarker discovery and validation study. Clin Epigenetics. 2019 Nov 14;11(1):158. doi: 10.1186/s13148-019-0757-3. PMID 31727158
- [Background] Jensen SO, Ogaard N, Nielsen HJ, Bramsen JB, Andersen CL. Enhanced Performance of DNA Methylation Markers by Simultaneous Measurement of Sense and Antisense DNA Strands after Cytosine Conversion. Clin Chem. 2020 Jul 1;66(7):925-933. doi: 10.1093/clinchem/hvaa100. PMID 32460325
- [Background] Ogaard N, Reinert T, Henriksen TV, Frydendahl A, Aagaard E, Orntoft MW, Larsen MO, Knudsen AR, Mortensen FV, Andersen CL. Tumour-agnostic circulating tumour DNA analysis for improved recurrence surveillance after resection of colorectal liver metastases: A prospective cohort study. Eur J Cancer. 2022 Mar;163:163-176. doi: 10.1016/j.ejca.2021.12.026. Epub 2022 Jan 22. PMID 35074652